CLINICAL TRIAL: NCT04284826
Title: The Clinical Efficacy of Endoscopic Postdilation Intralesional Injection of Mitomycin-C in Adults With Refractory Benign Esophageal Stricture
Brief Title: Mitomycin-C Injection Therapy in Refractory Esophageal Stricture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jin Hong Kim, Professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-MED-CT4-11-203
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Stricture
Keywords: Esophageal Stricture; mitomycin C; endoscopy
MeSH Terms: conditions — Esophageal Stenosis

STUDY DESIGN:
Intervention Model Description: Endoscopic intralesional Mitomycin-C injection in patients with refractory benign esophageal stricture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mitomycin C injection group (Experimental): A submucosal needle injection of 4mL of a MMC preparation (0.5mg/mL) into the tearing esophageal wall after esophageal bougie dilation on refractory benign esophageal stricture
  Interventions: Procedure: Endoscopic injection of Mitomycin-C on bougie-dilated refractory benign esophageal stricture

INTERVENTIONS:
Procedure: Endoscopic injection of Mitomycin-C on bougie-dilated refractory benign esophageal stricture

SUMMARY:
Intralesional Mitomycin-C (MMC) injection has recently been introduced to resolve refractory benign esophageal stricture mostly in children. The investigators aimed to evaluate the clinical efficacy of endoscopic postdilation intralesional injection of MMC in adults with refractory benign esophageal stricture.

DETAILED DESCRIPTION:
The participnts who have refractory benign esophageal stricture even after five or more sessions of bougination are prospectively enrolled. A submucosal needle injection of 4mL of a MMC preparation (0.5mg/mL) is endoscopically done with a 0.5mL of eight each injection mainly into the tearing esophageal wall, after esophageal bougie dilation is done upto 14mm in diameter. And then, repeated bouginations combined with MMC injection are done with the interval of eight weeks upto 3 times, if dysphagia symptoms recurr with dysphagis score 3 or more. Initial and overall clinical success rates are evaluated with drug and procedure-related complication rates during the follow-up period of at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 29 year and less than 75 year
* refractory benign esophageal stricture who had the symptoms of dysphagia score suggested by Mellow et al greater than 3 (0: able to eat a normal diet, 1: able to eat some solid food, 2: able to eat some semi-solids only, 3: able to swallow liquids only, 4: complete dysphagia)

Exclusion Criteria: Patients who have at least one of following conditions were excluded from our study

* malignant esophageal stricture
* multiple sites of esophageal stricture
* pregnant or breast feeding status
* clinical deterioration not tolerated to endoscopic procedures
* esophageal motility disorders
* esophageal leakage or fistula
* hypersensitivity to mitomycin C
* bleeding tendency due to thrombocytopenia or clotting disorders

Ages: 29 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Initial clinical success of mitomycin C injection therapy | 12 months after mitomycin C injection
  the improvement of dysphagia score more than one point after a single mitomycin C injection therapy during overall follow up period
Overall clinical success of mitomycin C injection therapy | 12 months after mitomycin C injection
  The improvement of dysphagia score more than one point after once or even after over twice mitomycin C injection therapy during follow up period

SECONDARY OUTCOMES:
Technical success of mitomycin C injection therapy | through study completion, an average of 1 year
  The successful performance of endoscopic mitomycin C injection into the submucosal layer at eight points of dilated stricture circumference after endoscopic dilation therapy
complications | through study completion, an average of 1 year
  endoscopic procedure-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hong Kim, Principal Investigator — Department of Gastroenterology, Ajou University School of Medicine, Suwon, Korea
Locations (1):
- Ajou University Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No